CLINICAL TRIAL: NCT07315204
Title: Viability Assessment Using Flavin Mononucleotide (FMN) Measured in Perfusate and Bile During Normothermic Machine Perfusion: an International, Multi-center Validation Study
Brief Title: Viability Assessment Using FMN Measured in Perfusate and Bile During Normothermic Machine Perfusion
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Andrea Schlegel, Director, Abdominal Transplant Research, The Cleveland Clinic
Other Study IDs: 25-839
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Liver Transplant Disorder
Keywords: normothermic machine perfusion; flavin mononucleotide; graft viability; liver transplant; OrganOx metra

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Recipients who receive deceased-donor liver transplant using machine perfusion with OrganOx metra: Normothermic perfusion using OrganOx metra. Can be from DBD or DCD donor.

SUMMARY:
Discarded perfusate samples will be collected from donors after circulatory death (DCD) or donors after brain death (DBD) organs during the machine perfusion period prior to transplantation by the study team. FMN will be measured as is standard of care for all machine perfusion liver transplant cases at Cleveland Clinic.

Participating centers will be provided with sample collection and shipping instructions to ensure sample preservation in accordance with IATA guidelines. Samples from outside sites will not be stored for future research and will be discarded once analysis is completed.

After the collection of the samples from machine perfusion, the transplant procedure will continue according to standard process.

DETAILED DESCRIPTION:
Real-time identification of graft viability is critical to safe expansion of the donor pool. Different strategies for viability testing in Normothermic Machine Perfusion (NMP) have been described by groups from the United Kingdom, The Netherlands, Austria, United States and Switzerland. In general, strategies in NMP utilize clinical observations, perfusion conditions, plus perfusate and bile analyses including lactate clearance, pH, glucose utilization/reuptake and more. At present there is no consensus for viability parameters or certain thresholds, though lactate clearance and clinical observation seem to be the most widely used criteria at present time.

Viability assessment has been reported for Hypothermic oxygenated perfusion (HOPE)-treated grafts, mostly centered around Flavin Mononucleotide (FMN), a marker of mitochondrial injury originating from mitochondrial Complex 1. FMN was shown to be released into perfusate at reoxygenation of previously ischemic tissues and correlating well with posttransplant complications and predicting graft loss beyond certain perfusate thresholds obtained during HOPE. This has led to improvements in graft loss and reduction of clinically relevant non-anastomotic strictures (NAS) with HOPE despite the use of extended criteria DCD livers (any donor age up to 100 years, old donors, >30min functional donor warm ischemia time (fDWIT), up to 8hrs static cold storage before HOPE, macrosteatosis) in Europe. Dr. Schlegel's group has recently validated prior thresholds center wide and internationally repeatedly showing the correlation between perfusate FMN and clinically relevant post-LT outcomes.

The investigators have investigated the utility of perfusate FMN obtained during NMP using the OrganOx metra device predicting graft loss and complications. Specifically, the investigators find that FMN predicts NAS, overall complications and graft loss after transplant. Perhaps most impressively, the investigators find that quantitative measurement of FMN can predict not only binary complications, but also severity of such complications in perfused grafts. The investigators further find that typical parameters such as lactate, glucose and bile chemistry are poorly correlated with post-transplant outcomes.

Finally, the investigators have validated FMN measured in bile as an add on identifying biliary injury in both a binary and a quantitative sense, specifically predicting biliary complications with different clinical severity and need for interventions.

This is a multicenter observational validation study. It is estimated 850 that patients will be needed across 10-15 study sites to confirm FMN as a viability marker during NMP. Around 250 patients will be enrolled from Cleveland Clinic, both retrospectively and prospectively, from October 22, 2022 - December 31, 2027.

- The primary aim of this study is to confirm and validate the ability of Flavin Mononucleotide (FMN) as a marker of future graft viability. The investigators aim in total for 10 to 15 participating centers, both in the US and UK, utilizing back-to-base normothermic machine perfusion with the OrganOx metra device.

Primary Endpoint: Graft functionality up to 1-year post-transplant, as measured by perfusate FMN, bile FMN and perfusate + bile FMN correlation with graft viability (Primary Non-function (PNF), non-anastomotic stricture (NAS), other related graft loss - death censored).

Secondary Endpoints:

* Clinically significant non-anastomotic strictures (NAS requiring intervention).
* All biliary complications, including AS, NAS, bile leaks
* Clinically significant NAS leading to graft loss
* Number of interventions required per NAS
* Complications according to Clavien-Dindo grading and comprehensive Complications Index (CCI)
* Primary nonfunction (PNF), early allograft dysfunction (EAD)
* Hepatic artery thrombosis (HAT) and other vascular complications
* Acute kidney injury (AKI), renal replacement therapy (RRT)
* Acute cellular rejection, number of biopsies, number of rejection episodes and severity
* Graft loss, death censored graft loss, recipient death, times and causes

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Any graft type (DBD or DCD)
* Any underlying recipient disease (i.e., end stage, liver tumour)
* Any other donor risk factors and static cold storage time prior to NMP accepted by the participating center for transplantation in context of OrganOx metra use
* Patients undergoing primary deceased donor liver transplantation where back-to-base NMP is used (OrganOx metra) from July 15, 2025 to December 31, 2027. (CCF only)
* Patients who have undergone deceased donor liver transplantation where back-to-base NMP was used (OrganOx metra) from October 22, 2022 to July 14, 2025. (CCF only)

Exclusion Criteria:

* Patients receiving a liver graft that is not perfused with OrganOx metra
* Pediatric recipients (<18years)
* Patients listed for super urgent liver transplantation due to acute liver failure
* Patients receiving combined organ transplant (heart+liver, lung+liver, liver+kidney, liver+intestine)
* Patients receiving living donor liver transplant or a split (or reduced) liver transplantation or a domino graft.
* Re-transplantations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recipients of deceased-donor liver transplant (DCD and DBD) will be recruited from outpatient clinics and inpatient services at the Cleveland Clinic Foundation Main Campus in the department of liver transplant. Patients will undergo their complete liver transplant work-up as directed by the multi-disciplinary selection committee and under the national direction of the United Network for Organ Sharing (UNOS). After completing their work-up, patients are discussed at the Liver Transplant Selection Committee, who must come to a consensus agreement regarding a candidate's eligibility prior to transplant. Each patient undergoing primary liver transplantation alone for end stage liver disease and/or liver tumor is eligible once approved by the committee, because this is an observational study comparing perfusion samples with standard-of-care clinical outcomes.
  Participating centers in this study will follow the standard procedures of their respective institutions.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Graft functionality as measured by FMN correlation with graft viability at 1 year post transplant | 1 year post transplant
  Graft functionality measured by perfusate FMN, bile FMN, and perfusate + bile FMN. Graft viability measured by primary non-function (PNF). Non-anastomotic stricture (NAS), other graft related loss - death censored.

SECONDARY OUTCOMES:
Clinically significant non-anastomotic strictures | within 1 year post-transplant
  Number of non-anastomotic strictures requiring intervention
Number/percentage of biliary complications | within 1 year post-transplant
  Biliary complications include anastomotic stricture (AS), NAS, bile leaks, as seen on imaging, ERCP/MRCP.
Clinically significant NAS leading to graft loss | within 1 year post-transplant
  Number of non-anastomotic strictures that result in graft failure
Number of interventions required per NAS | within 1 year post-transplant
Number of complications according to Clavien-Dindo grading and comprehensive Complications Index (CCI) | within 1 year post-transplant
Percentage of patients with primary nonfunction (PNF) and early allograft dysfunction (EAD) | within 7-10 days post-transplant
  EAD defined using Olthoff Criteria. PNF defined as non-functioning liver with patent vessels with 7 days after liver transplant.
Percentage of subjects with hepatic artery thrombosis (HAT) and other vascular complications | within 1 year post-transplant
  Subjects will be followed from time of surgery for at least one year post-transplant per institute standard. Complications, surgeries, etc will be collected and analyzed.
Number/Percentage of subjects with acute kidney injury (AKI), renal replacement therapy (RRT) | within 1 year post-transplant
Number/percentage of subjects with acute cellular rejection (ACR) | within 1 year post-transplant
  For subjects with ACR, the number of biopsies, number of rejection episodes, and the severity will be reported
Graft loss | within 1 year post-transplant.
  Number of grafts lost. Death censored graft loss, number of patient deaths, times, and causes of death.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Schlegel, MD, MBA, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No